CLINICAL TRIAL: NCT06163482
Title: Changes in Postprandial Hormone Levels in Cystic Fibrosis Related Diabetes.
Brief Title: Hormonal Responses to a Mixed Meal in People With Cystic Fibrosis
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Jason Winnick, Principal Investigator, University of Cincinnati
Other Study IDs: 2022-0593
Record Dates: First submitted 2023-11-27; First posted 2023-12-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
Keywords: diabetes; cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Human plasma samples will be analyzed for substrates and hormones.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy controls: No cystic fibrosis (CF)
  Interventions: Other: Mixed meal
- Pancreatic sufficient CF: cystic fibrosis, but not pancreatic insufficient
  Interventions: Other: Mixed meal
- Pancreatic insufficient CF: cystic fibrosis and pancreatic insufficient
  Interventions: Other: Mixed meal
- CF-related diabetes: cystic fibrosis and diabetes
  Interventions: Other: Mixed meal

INTERVENTIONS:
Other: Mixed meal — Each individual will ingest 5 mL/kg of Boost energy drink.

SUMMARY:
In this exploratory study, the hormonal responses to a mixed meal will be examined in people with cystic fibrosis. The aim of this study is to find correlates with impaired glucose tolerance that is associated with this population.

DETAILED DESCRIPTION:
The pancreas plays a key role in the regulation of whole-body glucose metabolism in humans. It contains 1 to 3 million islets, each of which contains several types of endocrine cells including insulin-secreting beta cells, glucagon-secreting alpha cells, and somatostatin- secreting delta cells. Insulin is released in response to a rise in blood glucose after a meal, and promotes glucose utilization by peripheral tissues (e.g., skeletal muscle), which allows the return of blood glucose to a fasting level. Glucagon is released when blood glucose falls below a normal fasting level (~80-100 mg/dL) and it acts on the liver in opposition to insulin, enhancing hepatic glucose production. Somatostatin's role in whole body glucose homeostasis is somewhat more complex. The role it plays in acutely regulating whole-body glucose homeostasis is small in healthy humans. On the other hand, it is capable of inhibiting the secretion of both insulin and glucagon, regardless of ambient metabolic conditions. In addition to its ability to regulate hormone secretion, somatostatin is also known to reduce glucose absorption from the gastrointestinal tract.

CF is the most common life-limiting genetic disease in Caucasians. It is caused by recessive mutations in the gene encoding CF transmembrane conductance regulator (CFTR). The primary pathologic change is secretion of thick ductular mucus, which leads to progressive obstructive damage to the lungs and exocrine pancreas. Damage to the exocrine pancreas, which is responsible for the secretion of digestive enzymes, leads to exocrine pancreas insufficiency (PI) manifested as diarrhea and malabsorption of ingested nutrients, requiring pancreatic enzyme replacement. Pathological changes of exocrine PI occur as early as the first few months of life, and most CF patients are diagnosed with PI before they reach adulthood.

The degree of exocrine PI correlates with risk of developing cystic fibrosis related diabetes (CFRD). However, not all CF patients with PI have diabetes. Patients with CFRD have impaired pancreatic beta cell function which is characterized most prominently by a loss of insulin secretion in response to the ingestion of glucose. Furthermore, it has been reported that glucagon responses to insulin induced hypoglycemia are reduced in CFRD, thereby providing evidence that pancreatic alpha cell function is also impaired in CFRD. One hypothesis for impaired endocrine function in CFRD is a reduction in islet count and/or altered islet-structure. These changes, which are hallmark characteristics of CF, are thought to be preceded by obstructive damage to the exocrine pancreas by thick, viscous pancreatic secretions that result in progressive fibrosis and fatty infiltration of the pancreas. Indeed, immunohistochemical studies of islets from patients with CFRD show significantly reduced insulin-producing cells compared to those of CF patients without diabetes and controls.

It is clear that metabolic regulation becomes progressively worse as the CF phenotype progresses from mild to severe (from exocrine pancreatic sufficiency, to exocrine pancreatic insufficiency, to diabetes). However, the mechanism through which this worsening of metabolic regulation occurs is unclear. In fact, it is possible that in addition to changes in islet morphology, another important factor that could lead to deteriorating metabolic regulation in CF is the mucosal secretions that result in fibrosis and fat infiltration in the pancreas. The aim of the current study is to examine how hormone responses to a mixed meal differ between healthy controls and people with cystic fibrosis, and how these changes correlate with deteriorating glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cystic fibrosis
* Aged 18 to 45 years
* Males and females of any race and ethnicity
* Receiving highly effective CFTR modular therapy

Exclusion Criteria:

* Transplant recipient
* Acute lung function decline or exacerbation within the last 3 months
* Use of systemic glucocorticoids
* Pregnancy
* Known liver disease that would be expected to significantly impact metabolic variable as interpreted by a study doctor
* The presence of any other disease or condition, as interpreted by any one of the study doctors, that would be expected to confound the responses to liquid mixed meal or make participation in the study dangerous to the individual
* People who are cognitively impaired
* People who do not speak English
* For CFRD patients, a daily insulin requirement that exceeds 0.8 U/kg/day
* Any prior history of diabetic ketoacidosis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy controls and people with cystic fibrosis will be examined.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of Insulin | Up to 3 hours
  human plasma
Concentration of Glucagon | Up to 3 hours
  human plasma
Concentration of Somatostatin | Up to 3 hours
  human plasma
Concentration of Glucose | Up to 3 hours
  human plasma

SECONDARY OUTCOMES:
Concentration of GLP-1 | Up to 3 hours
  human plasma
Concentration of GIP | Up to 3 hours
  human plasma
Concentration of fatty acids | Up to 3 hours
  human plasma

CONTACTS AND LOCATIONS:
Overall Officials: Jason Winnick, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No